CLINICAL TRIAL: NCT00675688
Title: A Double-Blind, Randomized, Placebo- and Active-Controlled Safety and Efficacy Study of Bazedoxifene/Conjugated Estrogens Combinations in Postmenopausal Women
Brief Title: Study Evaluating Safety and Efficacy of Bazedoxifene/Conjugated Estrogens Combinations in Postmenopausal Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3115A1-303
Record Dates: First submitted 2008-05-07; First posted 2008-05-12 (Estimated); Last update posted 2008-05-12 (Estimated); Status verified 2008-05

CONDITIONS: Endometrial Hyperplasia; Osteoporosis
Keywords: Menopause
MeSH Terms: conditions — Endometrial Hyperplasia; Osteoporosis | interventions — bazedoxifene; Raloxifene Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental)
  Interventions: Drug: Bazedoxifene/Conjugate Estrogens (CE)
- B (Active Comparator)
  Interventions: Drug: Raloxifene
- C (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bazedoxifene/Conjugate Estrogens (CE)
  Arms: A
Drug: Raloxifene
  Arms: B
Drug: Placebo
  Arms: C

SUMMARY:
The purpose of this study is to determine whether bazedoxifene/conjugated estrogens combinations are effective for the prevention of endometrial hyperplasia and for the prevention of osteoporosis in postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy, postmenopausal women aged 40 - 75 years inclusive
* Intact uterus
* Last natural menstrual cycle (without exogenous hormone therapy) completed at least 12 consecutive months before screening

Exclusion Criteria:

* A history or active presence of thrombophlebitis, thrombosis or thromboembolic disorders
* A history or active presence of cerebrovascular accident, stroke, or transient ischemic attack
* A history or active presence of malignancy, or treatment for malignancy, within the previous 10 years

Additional criteria applies.

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3544 (Actual)
Dates: Start 2002-04; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the effects of Bazedoxifene/Conjugate Estrogens (CE) combinations on the incidence of endometrial hyperplasia in postmenopausal women. | one year

SECONDARY OUTCOMES:
To evaluate the efficacy of Bazedoxifene/CE combinations in preventing osteoporosis. To evaluate the effects of Bazedoxifene/CE combinations on vaginal atrophy, metabolic parameters, uterine bleeding, vasomotor symptoms and quality of life indices. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer

REFERENCES:
- [Derived] Archer DF, Freeman EW, Komm BS, Ryan KA, Yu CR, Mirkin S, Pinkerton JV. Pooled Analysis of the Effects of Conjugated Estrogens/Bazedoxifene on Vasomotor Symptoms in the Selective Estrogens, Menopause, and Response to Therapy Trials. J Womens Health (Larchmt). 2016 Nov;25(11):1102-1111. doi: 10.1089/jwh.2015.5558. Epub 2016 Sep 27. PMID 27676118
- [Derived] Lobo RA, Pinkerton JV, Gass MLS, Dorin MH, Ronkin S, Pickar JH, Constantine G. Evaluation of bazedoxifene/conjugated estrogens for the treatment of menopausal symptoms and effects on metabolic parameters and overall safety profile. Fertil Steril. 2009 Sep;92(3):1025-1038. doi: 10.1016/j.fertnstert.2009.03.113. Epub 2009 Jul 26. PMID 19635615